CLINICAL TRIAL: NCT04853056
Title: The Effect of Virtual Reality and Cold Vibration Device on First Attempt Success, Procedure-Related Fear, Anxiety and Pain During Pediatric Intravenous Line Placement in Children Between 4-10 Years Old in the Emergency Department
Brief Title: Virtual-Reality and Cold-Vibration Device on Procedure-Related Fear, Anxiety and Pain During Pediatric IV Line Placement
Acronym: IVVRBuzzy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: xxx-GOA
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Pain; Fear; Anxiety; Child, Only
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Virtual Reality Group (Experimental): watching the application by wearing virtual glasses to the child during the peripheral IV line insertion
  Interventions: Device: virtual reality
- Cold Vibration Group (Experimental): Buzzy, connecting and operating 5 cm above the area to be inserted peripheral IV line
  Interventions: Device: Cold vibration
- Control group (No Intervention): Standart care

INTERVENTIONS:
Device: virtual reality — wearing virtual reality glasses
  Other Names: distraction methods
  Arms: Virtual Reality Group
Device: Cold vibration — Buzzy
  Other Names: distraction methods
  Arms: Cold Vibration Group

SUMMARY:
Studies evaluating VR are quite insufficient. In the study we determined in the emergency room between the ages of 4-10, cold vibration and virtual reality will be compared, and the success of the first attempt, pain, fear and anxiety will be evaluated.

DETAILED DESCRIPTION:
It was planned to evaluate the effect of virtual reality, cold vibration device application on the first attempt success, procedure-related pain, fear and anxiety during pediatric intravenous line placement in children aged 4-10 years in the pediatric emergency unit.

H1: Patients who watch videos with virtual reality glasses or who are applied cold vibration device during the vascular access procedure have a high first-attempt success.

H2: The pain, fear, and anxiety scores of the patients who watch videos with virtual reality glasses or who are applied cold vibration device during the venipuncture procedure are lower.

It is planned to include children between the ages of 4 and 10 who will be given vascular access in the Dokuz Eylül University Pediatric Emergency Unit. Between December 2020 and January 2021, it is planned to include patients selected by stratified randomization method in accordance with the sampling criteria. In the Gpower statistical program, based on the results of one-way variance analysis used in the comparison of pain and anxiety scores in the study of Canbulat et al. It was determined that a sample was required. In the study, it was planned to fulfill the parametric test assumptions and to have 50 children for each group and 150 children for the total sample, considering 10% loss.

Inclusion / exclusion criteria in the study:

* Children between the ages of 4-10
* The child agrees to voluntarily participate in the study.
* Parents agree to voluntarily participate in the study
* Obtaining consent form from the child and parent
* The child does not have a physical and psychological deficit to prevent him from wearing the glasses to be worn on his head so that he can watch virtual reality.

Patients who will be peripheral IV line accessed will be allocated to the groups according to randomization. The child and parents will be informed and after their consent, the group they belong to will be determined. No additional intervention will be made to the patient in the control group and will be observed during the procedure after obtaining her consent.

Standard approach will be applied to all pediatric patients. Standard approach; Providing information about the procedure, introducing the nurse himself, choosing the region together, being with the parent and talking to the child during the procedure. No additional intervention will be made to the patient in the control group, and until the intervention begins, "How old are you? Which grade are you in? What is the name of your favorite friend? Which sport do you like better? " Attention will be distracted by asking questions such as.

By introducing a virtual headset to the selected child to the video monitoring initiative group with virtual glasses, it will be said that he can watch videos by wearing the virtual headset during the procedure (Figure 1). The video he wants to watch together will be determined. If virtual glasses are desired to be removed during the procedure, the child will be excluded from the study. One of the 3 interesting videos will be determined by the researchers, with the preference of the child.

In the cold vibration group, bee Buzzy will be attached to the arm where the nurse will perform the peripheral IV line access. Bee Buzzy confuses nerves and reduces pain thanks to its cold wings and vibration. help distract attention during the injection period, reduce the feeling of pain and fear. Buzzy will be tied 5 cm above the area where blood will be taken, and after waiting 15 seconds, vascular access will be opened by the nurse. It will be wiped with disinfectant before and after the intervention.

After each patient included in the study is taken to the chair where the intervention will be performed (the starting hour/minute of the procedure will be recorded), the patient will be monitored and pulse, respiration, and blood pressure will be measured. The child will be evaluated by the nurse before the procedure with the Emotional Appearance Scale for Children.

The patient's pulse, respiration, blood pressure will be measured again (minutes will be recorded). Pulse, respiration and blood pressure will be re-evaluated at the 5th minute of the beginning of the procedure. At the 5th minute of the procedure, the child will be asked to evaluate the most painful moment he feels during the procedure with a Facial Expressions Rating Scale and a Color Analog Scale. The child will be given the Child Fear Scale (CFS) and the Child Anxiety Scale-State to evaluate how anxious and afraid he or she is during the procedure. You will be asked to mark it with a pencil.

Research data will be collected by the following data collection forms:

Socio-Demographic Data Collection Form Procedure Follow-up Form Pain scale Fear Scale Child Anxiety Scale-State Emotional Appearance Scale for Children

Socio-Demographic Data Collection Form: The Socio-demographic Data Collection Form consists of questions about the sociodemographic characteristics of the children and parents who will participate in the study. Sociodemographic features; It includes "age, gender, diagnosis, date of last bloodletting" regarding the child, and "age, closeness to the child, educational status, number of children" for the parent.

Procedure Follow-up Form: The child's difficult vascular access intervention score, procedure initiation time, vital signs, and first attempt success will be recorded.

Wong-Baker FACES (WBS) Pain Rating Scale. This scale uses in children aged 3 and older to rate pain severity, ranges from 0 (very happy/no pain) to 10 (hurts worst).

The Child Fear Scale (CFS). The Child Fear Scale will use.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear. This rating scale ranges from 0 to 4. It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome. The rater response indicates the level of fear. It can be used during the procedure for children aged 5-10 years.

The Children's Anxiety Meter (CAM-S). The Children's Anxiety Meter assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety.

Emotional Appearance Scale for Children: This scale allows direct behavioral observation, consists of 5 different behavioral categories; 'Facial Expression', 'Speaking', 'Activity', 'Interaction' and 'Cooperation Level'. Scale scoring is done by reviewing the descriptions of behavior in each category and selecting the numerical value that most represents the observed behavior. Each category is scored from 1 to 5. The total score is made so that the numerical value is between 5-25 by adding the points obtained for each category. Higher scale score indicates the appearance of more negative emotional behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 4-10
* The child agrees to voluntarily participate in the study.
* Parents agree to voluntarily participate in the study
* Obtaining consent form from the child and parent

Exclusion Criteria:

* - The child with physical and psychological deficit to prevent him from wearing the glasses to be worn on his head so that he can watch virtual reality.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Pain assesed by Wong-Baker FACES | during the procedure
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
Anxiety assesed by Children Anxiety Meter-State | during the procedure
  The Children's Anxiety Meter (CAM-S). The Children's Anxiety Meter assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety
Fear assesed by Child Fear Scale | during the procedure
  The Child Fear Scale (CFS). The Child Fear Scale will use.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear. This rating scale ranges from 0 to 4. It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome. The rater responds indicates the level of fear. It can be used during the procedure for children aged 5-10 years.

SECONDARY OUTCOMES:
Emotional Appearance Scale for Children | Baseline (before the procedure)
  This scale allows direct behavioral observation, consists of 5 different behavioral categories; 'Facial Expression', 'Speaking', 'Activity', 'Interaction' and 'Cooperation Level'. Scale scoring is done by reviewing the descriptions of behavior in each category and selecting the numerical value that most represents the observed behavior. Each category is scored from 1 to 5. The total score is made so that the numerical value is between 5-25 by adding the points obtained for each category. Higher scale score indicates the appearance of more negative emotional behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, Principal Investigator — RN, PhD, Assoc. Prof.
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No